CLINICAL TRIAL: NCT06749834
Title: Intravenous Thrombolytic Therapy in Acute Ischemic Stroke Patients on New Oral Anticoagulants
Brief Title: Intravenous Thrombolysis and NOAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I-NOAC
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Intravenous thrombolysis; outcome; NOAC
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous thrombolysis (Experimental): Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Interventions: Drug: Intravenous thrombolysis
- Standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Intravenous thrombolysis — Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Arms: Intravenous thrombolysis

SUMMARY:
New oral anticoagulants (NOACs), including rivaroxaban, apixaban, dabigatran, and edoxaban, have become the first-line therapy for preventing ischemic stroke associated with non-valvular atrial fibrillation (NVAF). Despite the effectiveness of NOACs in preventing thromboembolic events, approximately 1% to 2% of patients taking NOACs experience an ischemic stroke annually. Intravenous thrombolysis is an important means of treating acute ischemic stroke (AIS). However, due to concerns about the risk of symptomatic intracranial hemorrhage (sICH) or other severe bleeding complications, current guidelines still consider the use of NOACs within 48 hours before symptom onset as a contraindication to intravenous thrombolysis. Epidemiological data suggest that this may result in up to 18% of AF patients being unable to receive intravenous thrombolysis when they have an AIS episode.

Previous animal experiments have shown that NOACs do not increase the risk of hemorrhagic transformation after intravenous thrombolysis. Pharmacokinetic studies have demonstrated that 24 to 48 hours after taking NOACs, the anti-Xa level in patients is relatively low (<0.5 U/mL). In recent years, multiple retrospective studies and meta-analyses have shown that prior use of NOACs does not increase the risk of sICH in AIS patients receiving intravenous thrombolysis, and there are no significant differences in functional outcomes at 3 months. With solid pharmacokinetic and retrospective clinical evidence to support, it is hypothesized that IVT are safe in IS-NOAC patient. The investigators hereby propose a prospective multicenter study to determine the efficacy and safety of IVT in acute IS-NOAC.

DETAILED DESCRIPTION:
In this prospective cohort study, the investigators aim to recruit consecutive IS-NOAC patients who met the inclusion criteria. The investigators sought to determine the safety and efficacy of IVT in acute ischemic stroke patients on NOACs. It is hypothesized that for IS-DOAC patients with the last intake of NOAC within 48 hours, IVT improved neurological outcomes with acceptable safety compared to a cohort of acute IS-NOAC patients excluded from IVT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical signs of acute ischemic stroke within 24 hours of onset or awakening with stroke (if within 24 hours from the midpoint of sleep). Patients with AIS within 4.5-24 hours of onset must meet the IVT inclusion criteria specified in the guideline
2. Patients with new oral anticoagulants usage within 4-48 hours of onset;
3. Patients ≥ 18 years old
4. Informed consent has been obtained depending on local ethics requirements.

Exclusion Criteria:

1. Intended to proceed to endovascular treatment
2. With APTT >40s
3. Pre-stroke mRS score > 2
4. Contraindications for IVT：

1) Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hematoma, etc.) 2) Previous history of intracranial hemorrhage 3) Severe head trauma or stroke history within the last 3 months 4) Intracranial tumors, giant intracranial aneurysms 5) Intracranial or spinal surgery within the recent 3 months 6) Major surgical procedures within the last 2 weeks 7) Gastrointestinal or urinary tract bleeding within the last 3 weeks 8) Active visceral bleeding 9) Aortic arch dissection 10) Arterial puncture in a site within the last 1 week that is not easy to compress and stop bleeding 11) Elevated blood pressure: Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg 12) Acute bleeding tendency, including platelet count < 100 × 10⁹/L or other conditions 13) Received low-molecular-weight heparin treatment within 24 hours 14) Oral anticoagulants (warfarin) with INR > 1.7 or PT > 15 s 15) Blood sugar < 2.8 or > 22.22 mmol/L 16) Head CT or MRI indicates large-area infarction (infarction area ≥ 1/3 of the middle cerebral artery supply area) (4) The judgment is left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Excellent recovery assessed by the ratio of modified Rankin Scale (mRS) score of 0-1 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
the change on the National Institute of Health stroke scale (NIHSS) score from baseline to 1 day | from baseline to 1 day
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Independent recovery assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
recovery assessed by modefied Rankin Scale (mRS) score | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
3-month mortality | 90 ± 7 days
  Hospitalization records or follow-up results
Presence of parenchymal hemorrhage (PH) | at day 1
  the presence of PH is defined according the standard from ECASS-2 study
Presence of symptomatic intracerebral hemorrhage (sICH) | at day 1
  the presence of sICH is defined according the standard from ECASS-2 study
Presence of hemorrhagic transformation | at day 1
  Presence of hemorrhagic transformation is defined according the standard from ECASS-2 study

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Hangzhou, Zhejiang
  - The First People's Hospital of Wenling, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Protecting the privacy of participants is a priority, and sharing IPD could potentially compromise this.